CLINICAL TRIAL: NCT01042717
Title: Mobilization Kinetics of Plerixafor and G-CSF in Patients With NHL and MM Undergoing Autologous Peripheral Blood Progenitor Cell Collection
Brief Title: Study of the Best Timing for Plerixafor in Autologous Hematopoietic Stem Cell Collection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi, Patricia, M.D. (Individual)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Patricia Shi, Assistant Professor, Hematology-Oncology, Shi, Patricia, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO # 09-0824
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Multiple Myeloma; Non-Hodgkins Lymphoma
Keywords: plerixafor; autologous transplantation; hematopoietic stem cell mobilization; multiple myeloma; non-Hodgkins lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plerixafor (Experimental): Plerixafor 16 hours
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor administered at 16 hours prior to apheresis
  Other Names: Mozobil

SUMMARY:
The purpose of this study is to determine whether it is safe and effective to collect peripheral blood hematopoietic stem cells 16 hours rather than the usual 11 hours after administration of plerixafor.

DETAILED DESCRIPTION:
The current FDA-approved timing for plerixafor is approximately 11 hours prior to apheresis. This is a logistical problem, since plerixafor should be administered by a health care provider, given the risk of hypotension with administration. The primary purpose of this study is, in autologous donors with non-Hodgkins lymphoma and multiple myeloma undergoing hematopoietic progenitor cell mobilization with plerixafor and G-CSF, to determine whether the dosing interval can be increased to 16 hours prior to apheresis. Patients will be admitted to a special clinical research center on the 4th day of G-CSF administration, where the peripheral blood CD34+ count will be measured every 2 hours after plerixafor administration at 5 pm until 9 AM the following day, at which time apheresis will commence. The hypothesis is that plerixafor administration 16 hours prior to apheresis is as safe and effective as plerixafor administration at 11 hours prior to apheresis.

ELIGIBILITY:
Inclusion Criteria:

1. Autologous donors age 18 to 75 years with NHL or MM scheduled to undergo peripheral blood stem cell collection as part of standard clinical care. Biopsy-confirmed diagnosis of NHL or MM is to have been done prior to the first mobilization.
2. In first or second CR or PR
3. ECOG performance status of 0 or 1
4. WBC count greater than 2.5 x 10e9/1
5. Absolute PMN count greater than 1.5 x 10e9/1
6. PLT count greater than 100 x 10e9/1
7. Serum creatinine less than or equal to 2.2 mg/dl
8. SGOT, SGPT, and total bilirubin less than 2.5 X upper limit of normal (ULN)
9. Cardiac and pulmonary status sufficient to undergo apheresis and transplantation
10. Negative for HIV
11. 4 weeks since last cycle of chemotherapy. (Rituximab, thalidomide, dexamethasone, and bortezomib are not considered chemotherapy for the purpose of the study)
12. Patients of childbearing potential agree to use an approved form of contraception
13. Recovered from all acute toxic effects of prior chemotherapy

Exclusion Criteria:

1. Comorbid condition which renders patient, in view of the investigators, at high risk of treatment complications
2. Failed previous stem cell collections or collection attempts
3. Less than 6 weeks of carmustine prior to the 1st dose of G-CSF
4. Received GM-CSF or pegfilgrastim within 3 weeks prior to the 1st dose of G-CSF for mobilization
5. Received G-CSF within 14 days prior to the 1st dose of G-CSF for mobilization
6. Active CNS involvement
7. Active brain metastases or carcinomatous meningitis
8. Bone marrow involvement greater than 20 percent
9. Received radiation therapy to the pelvis
10. Post-transplant chemotherapy and/or radiation therapy below the diaphragm is anticipated
11. Received prior radio-immunotherapy with Zevalin or Bexxar
12. Fever (temperature greater than 38 C/100.4 F)
13. Received bone-seeking radionuclides (e.g., holmium)
14. A residual acute medical condition resulting from prior chemotherapy
15. Active brain metastases or myelomatous meningitis
16. Received thalidomide, dexamethasone and/or Velcade within 7 days prior to the first dose of G-CSF
17. Received Revlimid within 3 weeks prior to the first dose of G-CSF
18. Received greater than 6 cycles of Revlimid
19. Positive pregnancy test or lactating
20. Active infection requiring antibiotic treatment
21. Abnormal ECG with clinically significant rhythm disturbance (ventricular arrhythmias), or other conduction abnormality in the last year that in the opinion of the investigator warrants exclusion of the subject from the trial.
22. Patients who previously received experimental therapy within 4 weeks of enrolling in this protocol or who are currently enrolled in another experimental protocol during the mobilization phase.
23. Patients whose apheresis product will be further selected and purified.
24. Prior autologous or allogeneic transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Percent of donors obtaining a minimum CD34+ cell dose of 2 x 106/kg actual recipient weight within 2 days of collection | After collection

SECONDARY OUTCOMES:
Median and average neutrophil and platelet engraftment | After stem cell infusion
Plerixafor-related toxicities | 1 month after stem cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Shi, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Liles WC, Rodger E, Broxmeyer HE, Dehner C, Badel K, Calandra G, Christensen J, Wood B, Price TH, Dale DC. Augmented mobilization and collection of CD34+ hematopoietic cells from normal human volunteers stimulated with granulocyte-colony-stimulating factor by single-dose administration of AMD3100, a CXCR4 antagonist. Transfusion. 2005 Mar;45(3):295-300. doi: 10.1111/j.1537-2995.2005.04222.x. PMID 15752146
- [Background] DiPersio JF, Micallef IN, Stiff PJ, Bolwell BJ, Maziarz RT, Jacobsen E, Nademanee A, McCarty J, Bridger G, Calandra G; 3101 Investigators. Phase III prospective randomized double-blind placebo-controlled trial of plerixafor plus granulocyte colony-stimulating factor compared with placebo plus granulocyte colony-stimulating factor for autologous stem-cell mobilization and transplantation for patients with non-Hodgkin's lymphoma. J Clin Oncol. 2009 Oct 1;27(28):4767-73. doi: 10.1200/JCO.2008.20.7209. Epub 2009 Aug 31. PMID 19720922
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a609018.html